CLINICAL TRIAL: NCT07149142
Title: Feasibility and Effectiveness of Diabetic Retinopathy Screening Using Artificial Intelligence in Children With Type 1 Diabetes
Brief Title: Pediatric Artificial Intelligence for Retinopathy Screening in Children With Type 1 Diabetes
Acronym: PAIRS-T1D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Vit Neuman, MD, PhD, University Hospital, Motol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PAIRS
Record Dates: First submitted 2025-08-14; First posted 2025-08-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetic Retinopathy; Diabetic Neuropathy; Artificial Intelligence
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Retinopathy; Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): All participants will undergo 3 consecutive examinations - non-mydriatic fundus camera assessed by AI-driven software, fundus opthalmoscopy assessed by experienced opthalmologist and optic coherence tomography examination.
  Interventions: Diagnostic Test: Non-mydriatic fundus camera photography; Diagnostic Test: Fundus ophtalmoscopy; Diagnostic Test: Optic coherence tomography; Diagnostic Test: Confocal microscopy of the retina

INTERVENTIONS:
Diagnostic Test: Non-mydriatic fundus camera photography — Non-mydriatic fundus camera photography assessed by artificial intelligence software
Diagnostic Test: Fundus ophtalmoscopy — Fundus opthalmoscopy assessed by an experienced ophtalmologist
Diagnostic Test: Optic coherence tomography — Optic coherence tomography assessed by an experienced ophtalmologist
Diagnostic Test: Confocal microscopy of the retina — In a subset of participants over 18 years of age, confocal microscopy of the retina will be performed to assess the presence of diabetic neuropathy

SUMMARY:
The proposed project is a clinical intervention trial testing the feasibility and effectiveness of diabetic retinopathy screening evaluated by artificial intelligence (AI) based software in children with type 1 diabetes (CwD). Another novel method, the confocal microscopy of the retina will be used to assess the early stages of diabetic neuropathy. In parallel, we aim to assess the prevalence of diabetic retinopathy and neuropathy in a well-controlled population of CwD at a tertiary diabetes care center.

Each participant will undergo an examination of diabetic retinopathy using the non-mydriatic fundus camera. The resulting photography will be evaluated by AI driven software. The participant will then follow this examinaton with fundus ophtalmoscopy in arteficial mydriasis as a standard method of diabetic retinopathy assessment. Another method, the optic coherence tomography (OCT), which is considered as the most sensitive method for diabetic retinopathy assessment, will be performed after that. The results of these methods will be compared to assess the sensitivity of each. The examination-satisfaction questionnaire will be given to the participants.

In subjects over 18 years, a confocal microscopy of the retina examination will be performed to assess the status of the corneal sub-basal nerve plexus and the presence of diabetic neuropathy will be noted.

The prevalence of diabetic retinopathy and neuropathy in this group of children with diabetes will be assessed based on the results.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed according to the ADA criteria
* Age over 11.0 years or duration of diabetes over 2 years
* Signed written informed consent by both the CwD and their parent/caregiver

Exclusion Criteria:

* Unwillingness to sign a written informed consent by both the CwD and their parent/caregiver

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of AI for retinopathy screening | Through study completion, on average 6 months.
  The primary objective of this study is to test whether performing the diabetic retinopathy screening using the non-mydriatic fundus camera with AI software is feasible. The exact outcome is the percent of participants who will agree to undergo the procedure and will obtain a valid result (either positive or negative).

SECONDARY OUTCOMES:
Examination satisfaction | Through study completion, on average 6 months.
  Participant and caregiver reported examination satisfaction assessed by a structured questionnaire on a Lickert scale from 1 to 5.
Prevalence of diabetic retinopathy | Through study completion, on average 6 months.
  Prevalence of diabetic retinopathy among CwD in a single center with favorable glucose control
Prevalence of diabetic neuropathy | Through study completion, on average 6 months.
  Prevalence of diabetic neuropathy in young people with diabetes (over 18 years) in a single center with favorable glucose control

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Motol, Prague, Prague 5, Czechia

IPD SHARING:
Plan to Share IPD: Undecided